CLINICAL TRIAL: NCT06106828
Title: A Phase III, Randomized, Double-Masked, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Satralizumab in Participants With Moderate-to-Severe Thyroid Eye Disease
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Satralizumab in Participants With Thyroid Eye Disease
Acronym: SatraGO-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP44729; 2023-503669-50-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Eye Disease
Keywords: TED
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — satralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Satralizumab (Experimental): In the Part I period, participants will receive satralizumab every 4 weeks (q4w) followed by proptosis response-based individualized treatment in Part II of the study.
  Interventions: Drug: Satralizumab
- Placebo (Placebo Comparator): In the part I period, participants will receive placebo q4w followed by proptosis response-based individualized treatment in part II of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Satralizumab — Satralizumab will be administered by SC injection.
  Arms: Satralizumab
Drug: Placebo — Placebo will be administered by SC injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, safety, pharmacokinetics, and pharmacodynamics of subcutaneous (SC) satralizumab, a recombinant, humanized anti-interleukin-6 (IL-6) receptor monoclonal antibody, in participants with thyroid eye disease (TED).

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of TED based on CAS

Exclusion Criteria:

* Decrease in CAS or proptosis of >≥ 2 points or ≥ 2 mm, respectively, in the study eye between Screening and Study Baseline (Day 1)
* Requiring immediate surgical ophthalmological intervention or planning corrective surgery or irradiation during the course of the study, in the judgment of the investigator
* Identified pre-existing ophthalmic disease that, in the judgment of the investigator, would preclude study participation or complicate interpretation of study results, including corneal decompensation unresponsive to medical management and including ophthalmic diseases that will likely require prohibited therapy during the study
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes an individual's safe participation in and completion of the study
* Pregnant or breastfeeding, or intention of becoming pregnant during the study or within 3 months after the final dose of satralizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving ≥ 2 millimetres (mm) Reduction in Proptosis From Baseline (Day 1) at Week 24 in the Study Eye | Baseline, Week 24
  Provided there is no deterioration of proptosis (≥ 2mm increase) in the fellow eye.

SECONDARY OUTCOMES:
Change in Proptosis | Baseline, Week 24, Week 48, and from Week 24 to Week 48
Percentage of Participants Achieving ≥ 1 Grade Reduction/Improvement in Diplopia Among Participants With Baseline Diplopia | Baseline, Week 24, and Week 48
Percentage of Participants Achieving Absence of Motility-induced Pain | Week 24
Percentage of Participants Achieving Absence of Spontaneous Pain | Week 24
Percentage of Participants With a ≥ 6-Point Improvement in the Visual Functioning and Appearance Sub-scale Scores of the Graves' Ophthalmopathy Quality of Life (GO-QoL) | Baseline, Week 24, Week 48 and from Week 24 to Week 48
  The GO-QoL is a 16-item self-administered questionnaire divided into two sub-scales and used to assess the perceived effects of TED by the participants on their: 1) Visual Functioning (questions 1-8); and 2) Appearance (questions 9-16). Both the subscales and overall score are transformed to a scale of 0 to 100. Higher total scores indicate better QoL.
Percentage of Participants Achieving Overall Response | Week 24, Week 48
Percentage of Participants Achieving a ≥ 2 Point Reduction in Clinical Activity Score (CAS) in the Study Eye | Baseline, Week 24, and Week 48
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to TED; 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active TED (ignore "equivocal" redness); 6. Chemosis; 7. Swelling of caruncle or plica. Each item is scored as 1 (present) or 0 (absent) and scores for each item are summed for total score of 0 (no inflammatory symptoms) to 7 (most inflammatory symptoms). Higher scores indicate worse symptoms.
Percentage of Participants Achieving CAS Value of 0 or 1 in the Study eye | Week 24
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to TED; 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active TED (ignore "equivocal" redness); 6. Chemosis; 7. Swelling of caruncle or plica. Each item is scored as 1 (present) or 0 (absent) and scores for each item are summed for total score of 0 (no inflammatory symptoms) to 7 (most inflammatory symptoms). Higher scores indicate worse symptoms.
Percentage of Participants Achieving ≥ 10-point Improvement in Ocular Surface Disease Index (OSDI) Overall Scores | Baseline, Week 24
  The OSDI instrument is a validated dry eye questionnaire, designed to assess cornea and ocular surface symptoms. It comprises of 12 questions with three main sections concerning ocular symptoms, visual function, and environmental factors. For each question, participants selects a number between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time" with totals ranging from 0 to 100. Higher score indicates worse disease index.
Change in OSDI Ocular Symptoms and Vision-related Function Subscale Scores | Baseline, Week 24
  The OSDI instrument is a validated dry eye questionnaire, designed to assess cornea and ocular surface symptoms. It comprises of 12 questions with three main sections concerning ocular symptoms, visual function, and environmental factors. For each question, participants selects a number between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time" with totals ranging from 0 to 100. Higher score indicates worse disease index.
Change in Oxford Corneal Staining Scores | Baseline, Week 24
  Oxford corneal staining chart consists of a 6 point scale. Staining assessment will be based on the intensity of fluorescein staining, ranging from Grade 0 to V for each panel (Grade 0-I: normal; Grade II-III: mild to moderate; Grade IV-V: severe). Higher grade indicates worse disease index.
Percentage of Participants Achieving ≥ 2mm Reduction in Proptosis at Week 48 in the Study eye | Week 48
Percentage of Participants Requiring Surgical Intervention for TED | Up to Week 48
Percentage of Participants With Worsening of Proptosis by ≥ 2 mm | Baseline, Week 48 and from Week 24 to Week 48
Change in CAS | Baseline, Week 48 and from Week 24 to Week 48
Percentage of Participants With Adverse Events (AEs), With Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5 (NCI CTCAE V5) | Baseline up to Week 72
Serum Concentration of Satralizumab | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- United States (6):
  - Plastics-Orbit-Neuro, San Diego, California
  - Connecticut Eye Consultants, P.C., Danbury, Connecticut
  - University of Illinois Eye and Ear Infirmary, Chicago, Illinois
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Retina Consultants of Texas, San Antonio, Texas
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Toronto Retina Institute, Toronto, Ontario
  - Universite de Montreal - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- China (5):
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Hospital of Ministry of Health, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Xi'an Fourth Hospital, Xi'an
- France (3):
  - CHU Nantes - Hotel Dieu, Nantes
  - CHNO Hopital des Quinze Vingts, Paris
  - Fondation Rothschild, Paris
- Israel (3):
  - Hadassah MC, Jerusalem
  - Rabin MC, Petah Tikva
  - Sheba medical center, Ramat Gan
- Poland (2):
  - Specjalistyczny O?rodek Okulistyczny Oculomedica, Bydgoszcz
  - Profesorskie Centrum Medyczne Spolka Z Ograniczona Odpowiedzialnoscia, Gdansk
- AIBILI - Association for Innovation and Biomedical Research on Light, Coimbra, Portugal
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Chung-Ang University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario la Fe: Servicio de Oftalmologia, Valencia
- United Kingdom (7):
  - Sussex Eye Hospital, Brighton
  - Bristol Eye Hospital, Bristol
  - Gartnavel General Hospital, Glasgow
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Maidstone Hospital, Maidstone, Kent

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Ezra D, Collins A, Haskova Z, Kuenzel T, Ida H, Triyatni M, Brittain C, Idowu O. Targeting IL-6 Receptor Signaling with Satralizumab in Thyroid Eye Disease: Design of the Phase 3 SatraGO-1 and SatraGO-2 Trials. Ophthalmol Ther. 2025 Dec;14(12):3119-3132. doi: 10.1007/s40123-025-01255-3. Epub 2025 Oct 9. PMID 41066062